CLINICAL TRIAL: NCT04240314
Title: Phase I/IIa Systemic Gene Delivery Clinical Trial of scAAV9.U7.ACCA for Exon 2 Duplication-Associated Duchenne Muscular Dystrophy
Brief Title: AAV9 U7snRNA Gene Therapy to Treat Boys With DMD Exon 2 Duplications.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Megan Waldrop (Other)
Collaborators: Audentes Therapeutics (Industry); Astellas Pharma Inc (Industry)
Responsible Party: Sponsor-Investigator, Megan Waldrop, Professor of Neurology, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAV9 Dup2 U7
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Results first posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Intervention Model Description: This trial will deliver the minimal efficacious dose as determined by preclinical studies and approved by the FDA to determine safety and target engagement.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cohort 1 (Minimal Efficacious Dose) (Experimental): The Minimal Effective Dose (MED) will be delivered.
  Interventions: Biological: scAAV9.U7.ACCA

INTERVENTIONS:
Biological: scAAV9.U7.ACCA — A single dose of scAAV9.U7.ACCA will be systemically delivered via a peripheral vein injection.

SUMMARY:
Open-label, single dose clinical trial of scAAV9.U7.ACCA via peripheral limb vein injection for Duchenne muscular dystrophy boys who have a duplication of exon 2.

DETAILED DESCRIPTION:
The proposed clinical trial is a systemic (intravenous) delivery of scAAV9.U7.ACCA for DMD patients with a duplication of exon 2 in the DMD gene. Preclinical data shows that the small nuclear RNA (snRNA) construct delivered by the scAAV9.U7.ACCA vector causes significant skipping of exon 2, resulting in exclusion of the exon from the mature messenger RNA (mRNA) with a high degree of efficiency, leading to mRNA containing only a single exon 2 (wild type [WT] mRNA) or no copies of exon 2 (Del2 mRNA). Translation of the wild-type mRNA results in entirely normal dystrophin protein, whereas translation of the Del2 mRNA via translational initiation of an internal ribosome entry sequence, or IRES) results in a highly functional isoform expressed in patients known to walk into their eighth decade.

The study is designed as an open-label trial to assess safety and obtain preliminary efficacy data. scAAV9.U7.ACCA will be delivered to the systemic circulation via peripheral limb vein.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 6 months and less than 14 years
* Confirmed duplication of exon 2 in the DMD gene using a clinically accepted technique that completely defines the mutation
* Pre-ambulant (not yet walking) or ambulant (as defined by the ability to walk 10 meters without assistance)
* Males of any ethnic group will be eligible
* Ability to cooperate with muscle testing
* In subjects age 4 and above, stable dose and regimen of corticosteroid therapy (prednisone, deflazacort, or their generic forms) for at least 12 weeks prior to gene transfer.

Exclusion Criteria:

* Active viral infection based on clinical observations
* Symptoms or signs of cardiomyopathy, including:

  1. Dyspnea on exertion, pedal edema, shortness of breath upon lying flat, or rales at the base of the lungs
  2. Echocardiogram with ejection fraction below 40%
* Serological evidence of HIV infection, or Hepatitis B or C infection
* Diagnosis of (or ongoing treatment for) an autoimmune disease
* Persistent leukopenia or leukocytosis (WBC ≤ 3.5 K/µL or ≥ 20.0 K/µL) or an absolute neutrophil count < 1.5K/µL
* Concomitant illness or requirement for chronic drug treatment that in the opinion of the SI creates unnecessary risks for gene transfer
* AAV9 binding antibody titers ≥ 1:400 as determined by ELISA immunoassay
* Abnormal laboratory values in the clinically significant range as listed in Table 7, based upon normal values in the Nationwide Children's Hospital Laboratory.

Ages: 6 Months to 13 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 3 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2023-11-13 (Actual); Study Completion 2025-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Megan Waldrop, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Background] Wein N, Vulin A, Falzarano MS, Szigyarto CA, Maiti B, Findlay A, Heller KN, Uhlen M, Bakthavachalu B, Messina S, Vita G, Passarelli C, Brioschi S, Bovolenta M, Neri M, Gualandi F, Wilton SD, Rodino-Klapac LR, Yang L, Dunn DM, Schoenberg DR, Weiss RB, Howard MT, Ferlini A, Flanigan KM. Translation from a DMD exon 5 IRES results in a functional dystrophin isoform that attenuates dystrophinopathy in humans and mice. Nat Med. 2014 Sep;20(9):992-1000. doi: 10.1038/nm.3628. Epub 2014 Aug 10. PMID 25108525
- [Background] Vulin A, Wein N, Simmons TR, Rutherford AM, Findlay AR, Yurkoski JA, Kaminoh Y, Flanigan KM. The first exon duplication mouse model of Duchenne muscular dystrophy: A tool for therapeutic development. Neuromuscul Disord. 2015 Nov;25(11):827-34. doi: 10.1016/j.nmd.2015.08.005. Epub 2015 Aug 11. PMID 26365037
- [Background] Gurvich OL, Maiti B, Weiss RB, Aggarwal G, Howard MT, Flanigan KM. DMD exon 1 truncating point mutations: amelioration of phenotype by alternative translation initiation in exon 6. Hum Mutat. 2009 Apr;30(4):633-40. doi: 10.1002/humu.20913. PMID 19206170
- [Background] Flanigan KM, Dunn DM, von Niederhausern A, Howard MT, Mendell J, Connolly A, Saunders C, Modrcin A, Dasouki M, Comi GP, Del Bo R, Pickart A, Jacobson R, Finkel R, Medne L, Weiss RB. DMD Trp3X nonsense mutation associated with a founder effect in North American families with mild Becker muscular dystrophy. Neuromuscul Disord. 2009 Nov;19(11):743-8. doi: 10.1016/j.nmd.2009.08.010. Epub 2009 Sep 29. PMID 19793655
- [Background] Vulin A, Barthelemy I, Goyenvalle A, Thibaud JL, Beley C, Griffith G, Benchaouir R, le Hir M, Unterfinger Y, Lorain S, Dreyfus P, Voit T, Carlier P, Blot S, Garcia L. Muscle function recovery in golden retriever muscular dystrophy after AAV1-U7 exon skipping. Mol Ther. 2012 Nov;20(11):2120-33. doi: 10.1038/mt.2012.181. Epub 2012 Sep 11. PMID 22968479

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1 (Minimal Efficacious Dose)
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cohort 1 (Minimal Efficacious Dose)
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: Years] | 8 [0.7 to 14]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Unacceptable Toxicity.
Description: Unacceptable toxicity is defined as the occurrence of two or more unexpected Grade III or higher treatment-related toxicities, as defined by CTCAE 5.0.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Minimal Efficacious Dose)
Number analyzed (Participants) | 3
Participants | 0

2. Secondary Outcome: Change in Dystrophin Expression From Baseline Following Treatment With scAAV9.U7.ACCA.
Description: Expression of dystrophin will be measured by immunofluorescent (IF) staining in muscle biopsies taken before and after gene therapy. This method allows for visualization of the protein and its proper location in the muscle fiber in comparison to normal protein expression.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: % Change in dystrophin expression
Arm/Group | Cohort 1 (Minimal Efficacious Dose)
Number analyzed (Participants) | 3
% Change in dystrophin expression | 46.6 (36.8)

3. Secondary Outcome: Change in Dystrophin Expression From Baseline Following Treatment With scAAV9.U7.ACCA.
Description: Expression of dystrophin will be quantified by western blotting in muscle biopsies taken before and after gene therapy. This method allows for quantification of the protein amount in comparison to normal protein expression amounts.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: % Change in dystrophin expression
Arm/Group | Cohort 1 (Minimal Efficacious Dose)
Number analyzed (Participants) | 3
% Change in dystrophin expression | 30.1 (38.6)

4. Secondary Outcome: Changes in Percent of Exon 2 Skipping/Exclusion in the Dystrophin mRNA Transcript.
Description: Exon 2 exclusion will be measured using RT-PCR analysis.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: % Exon 2 Exclusion
Arm/Group | Cohort 1 (Minimal Efficacious Dose)
Number analyzed (Participants) | 3
% Exon 2 Exclusion
  Skipping of 1 Exon 2 | 4.9 (4.8)
  Skipping of 2 Exons 2 | 33.6 (45.4)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Cohort 1 (Minimal Efficacious Dose)
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (Minimal Efficacious Dose) (N=3)
Elevated ALT (Gastrointestinal disorders) | 1 (1)
Elevated AST (Gastrointestinal disorders) | 2 (4)
Hoarseness (Gastrointestinal disorders) | 1 (1)
Increased GI Reflux (Gastrointestinal disorders) | 2 (2)
Loose stool/Diarrhea (Gastrointestinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 3 (5)
Generalized Body Pain (General disorders) | 1 (1)
Irritability (General disorders) | 1 (1)
Mild to Moderate Dehydration (General disorders) | 1 (1)
Weight Gain (General disorders) | 1 (1)
COVID-19 Infection (Infections and infestations) | 3 (3)
Decreased ANC (Infections and infestations) | 1 (3)
Decreased Apetite (Infections and infestations) | 1 (1)
Decreased WBC (Infections and infestations) | 1 (1)
Fever (Infections and infestations) | 1 (2)
Right Great Toe Onychocyrptosis (Infections and infestations) | 1 (1)
Thrush (Infections and infestations) | 1 (1)
Viral Gastroenteritis (Infections and infestations) | 1 (1)
Viral Illness (URBX5, GI 5X5) (Infections and infestations) | 1 (1)
Viral Infection (Infections and infestations) | 1 (1)
Viral Syndrome (Infections and infestations) | 1 (1)
Decreased Vitamin D (Metabolism and nutrition disorders) | 1 (2)
Ankle Sprain (Musculoskeletal and connective tissue disorders) | 1 (1)
Right Heel Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Left foot discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Left Thigh Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Right Thing Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Upper and Midline Backpain (Musculoskeletal and connective tissue disorders) | 1 (1)
Erythematous Macuopapular Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Irritant Diaper Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Biopsy Site Discomfort (Surgical and medical procedures) | 2 (7)
Contact Dermatitis (Surgical and medical procedures) | 1 (2)
Flu-like Symptoms (Surgical and medical procedures) | 1 (1)
Left IV Site Pain (Surgical and medical procedures) | 1 (1)
Nausea (Surgical and medical procedures) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-18): https://cdn.clinicaltrials.gov/large-docs/14/NCT04240314/Prot_SAP_001.pdf